CLINICAL TRIAL: NCT00573066
Title: The Pharmacokinetics, Pharmacogenetics, and Pharmacodynamics of Dexmedetomidine In Infants Post-Operative From Cardiac Surgery
Brief Title: Understanding Dexmedetomidine In Infants Post-Operative From Cardiac Surgery
Acronym: InfantDex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athena Zuppa (Other)
Responsible Party: Sponsor-Investigator, Athena Zuppa, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-5-3770
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Hypoplastic Left Heart; Tetralogy of Fallot; Tricuspid Atresia
Keywords: Postoperative from cardiac surgery; Dexmedetomidine
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tetralogy of Fallot; Tricuspid Atresia | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dosing level (Experimental): A predetermined dose of Dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dosage levels: Dose Level 1: Loading dose 0.35mcg/kg and CIVI 0.25mcg/kg/hr Dose Level 2: Loading Dose of 0.7mcg/kg and CIVI 0.5mcg/kg/hr and Dose Level 3: Loading Dose 1 mcg/kg and CIVI 0.75 mcg/kg/hr.
  Other Names: Precedex

SUMMARY:
This study is being conducted to determine what dexmedetomidine does to the body and in turn, what how the body handles the medication. This medication, for the purpose of this trial, is used as a short-term sedative for infants who are immediately post-operative from cardiac surgery and have a breathing tube and are breathing with the assistance of a mechanical ventilator or breathing machine.

DETAILED DESCRIPTION:
This is a single center, dose escalation study of a single bolus dose of dexmedetomidine followed by a continuous infusion for up to 24 hours in infants who are immediately post-operative from cardiac surgery and require tracheal intubation with mechanical ventilation in the post-operative period. Three bolus doses and infusion doses will be administered to a total of 36 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater or equal to one month or less than or equal to 24 months of age.
* Post operative from cardiac surgery with tracheal intubation/mechanical ventilation in the immediate post-op period.
* Planned tracheal extubation within 24 hours post-operatively.
* Adequate renal function(1-12 months old creatinine less than or equal to 0.6mg/dL and >12 months to 24 months creatinine < or= to 1.0mg/dL)
* Adequate liver function(Total bilirubin < or= 1.5mg/dL and ALT 1-12 months < or = to 165 U/L and > 12 months to 24 months < or = to 90 U/L)
* Isolated heart surgery
* Informed consent

Exclusion Criteria:

* Patients who have received another investigational drug within the past 30 days.
* Receiving continuous infusions of muscle relaxants in the postoperative setting.
* Patients whoo have a positive blood culture without a subsequent negative culture or other evidence of ongoing serious infection.
* Patients, who, int he opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Patients who show signs or symptoms of elevated intracranial pressure.
* Post-operative hypotension based on age.
* Preexisting bradycardia based on age.
* Heart block
* Weight < 5kg
* Patients, who in the opinion of the investigator, are not appropriate candidates for an investigational drug study.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the CHOP cardiac center during preoperative evaluation.
Pre-assignment Details: All patients were evaluated postoperative to establish appropriateness for inclusion in the study.
Groups:
- Dexmedetomidine Dose Escalation Cohorts: Dexmedetomidine was administered to all subjects as an intravenous loading dose over 10 minutes followed by a continuous infusion for up to 24 hours.
  Cohort 1--0.35mcg/kg loading dose, 0.25mcg/kg/hr infusion Cohort 2--0.7 mcg/kg loading dose, 0.5 mcg/kg/hr infusion Cohort 3--1 mcg/kg loading dose, 0.75 mcg/kg/hr infusion
Period: Overall Study
Arm/Group | Dexmedetomidine Dose Escalation Cohorts
Started | 56
Completed | 36
Not Completed | 20
Not completed — Exclusion criteria | 18
Not completed — IV malfunction | 1
Not completed — Postoperative bleeding | 1

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine, Infants, Cardiac Surgery: Pharmacologic study of dexmedetomidine in infants following cardiac surgery Dexmedetomidine was administered to all subjects as an intravenous loading dose over 10 minutes followed by a continuous infusion for up to 24 hours.
  Cohort 1--0.35mcg/kg loading dose, 0.25mcg/kg/hr infusion Cohort 2--0.7 mcg/kg loading dose, 0.5 mcg/kg/hr infusion Cohort 3--1 mcg/kg loading dose, 0.75 mcg/kg/hr infusion
Arm/Group | Dexmedetomidine, Infants, Cardiac Surgery
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.74 (0.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: PK Profile of Dexmedetomidine
Description: This study measured the concentration of dex in the body and used those concentrations to determine how quickly the body metabolizes and eliminates dex(concentration-time or pharmacokinetic profile).The concentration of dex in the body is determined through serial blood sampling while administering dex and following discontinuation.
Time Frame: after start of infusion (0.5, 1, 2, 4-6 hours), immediately prior to end of infusion and following end of infusion (0.25, 0.5, 1, 2, 4, 8, 12, 15-18 hours)
Population: Based on an estimated inter-subject variability of 50% for steady state concentration, a sample size of 36 evaluable subjects will be sufficient to detect a difference (alpha 0.05, power 0.8) for the area under the concentration-time curve (AUC) and steady state concentration (Css) between the three dosing groups.
Measure: Least Squares Mean (Standard Error); unit: mL/min/(kg^0.75)
Arm/Group | Dexmedetomidine, Infants, Cardiac Surgery
Number analyzed (Participants) | 56
mL/min/(kg^0.75) | 28 (0.08)

ADVERSE EVENTS:
Time Frame: Data collected for up to 30 days following end of dexmedetomidine administration
Description: All adverse events possibly, probably and definitely related are included.
Arm/Group | Dexmedetomidine, Infants, Cardiac Surgery
Serious Adverse Events (participants affected / at risk) | 3/56
Other Adverse Events (participants affected / at risk) | 5/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine, Infants, Cardiac Surgery (N=56)
Hypotension (Cardiac disorders) | 2 (2) — Post-operative blood loss
Bradypnea/Oversedation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine, Infants, Cardiac Surgery (N=56)
Complete heart block (Cardiac disorders) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 3 (3)
Accelerated junctional rhythm (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No